CLINICAL TRIAL: NCT04977622
Title: Investigating Cortical Gray Matter Demyelination in Primary Progressive Multiple Sclerosis at 7 Tesla
Brief Title: Gray Matter Demyelination in Primary Progressive MS at 7T
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Scleroseforeningen (Unknown); Danish Multiple Sclerosis Center (Unknown)
Responsible Party: Principal Investigator, Hartwig R. Siebner, Professor, Danish Research Centre for Magnetic Resonance
Other Study IDs: A40219
Record Dates: First submitted 2021-04-06; First posted 2021-07-27 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Primary Progressive Multiple Sclerosis
Keywords: Magnetic Resonance Imaging; Ultra-high field MRI; Cortex; Multiple Sclerosis; Sensorimotor Function; Myelin; 7T; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Progressive MS (PPMS): Clinically definite MS patients with identified primary-progressive disease onset, within 10 years of diagnosis
- Non-neurological controls (HC): Age and sex matched to the PPMS patients

SUMMARY:
Progressive-onset multiple sclerosis (PPMS) occurs in about 15% of all people living with MS. PPMS remains understudied, and most disease-modifying treatments are ineffective for PPMS. To date, it is unknown why some people progress immediately from MS onset. The present study will assess the role of gray matter in PPMS by characterizing it with ultra-high field magnetic resonance imaging (MRI). While both white and gray matter are affected in relapsing MS, in PPMS tissue damage is primarily in the cortex. Cortical gray matter consists largely of neuronal cell bodies, which send electrical signals to create a functional response, such as arm or leg movement. While white matter damage slows the signal response, cortical damage inhibits the initial creation of electrical signals. There is a great need to research and develop scientific biomarkers to identify and monitor progression and repair in PPMS. In this project, 7 Tesla MRI is used to investigate the cortical gray matter in people with PPMS. 7 Tesla MRI is the safest and most detailed way to study the brain. Because the cortex is only a few millimeters thick, it has been traditionally difficult to investigate. At 7 Tesla, different layers and lesions within the cortex can be seen. In addition, this project will use myelin-sensitive MRI to determine the biological underpinnings of both cortical lesions and the 'normal appearing' cortical damage in PPMS. This will answer relevant questions about the brain's capacity for repair, the extent of demyelination and the occurrence of inherent cortical remyelination and provides an avenue for the development of novel clinical MR biomarkers tailored to PPMS.

DETAILED DESCRIPTION:
PURPOSE:

PPMS presents very differently from relapsing-remitting MS. Spinal cord involvement is greater and motor impairment significantly outweighs sensory symptoms. Contrast-enhancing lesions are infrequent in PPMS. Instead, gray matter atrophy and cortical demyelination occur at greater rates than in relapsing MS. Cortical involvement is prognostically relevant. MRI at standard clinical field strengths (e.g. 1.5 and 3 Tesla) has clear limitations for visualizing cortical damage. In particular, demyelination at the outer cortical layers is underestimated. Although 7 Tesla MRI is known to be superior to clinical MRI, myelin imaging has not yet been widely explored at 7 Tesla.

STUDY AIMS:

Use anatomical and quantitative MRI at 7 Tesla to identify radiologically visible and invisible features of cortical gray matter damage that contribute to physical and cognitive impairment in PPMS.

The specific project aims are

1. to utilize submillimeter anatomical MRI to map the distribution of the different types of cortical lesions in PPMS and assess cortical lesion volume and burden
2. to characterize and compare cortical lesions, perilesional gray and white matter as well as normal appearing gray matter (NAGM) using quantitative MR sequences
3. to explore the relationship between volumetric and myelin-measures with clinical scores in order to determine the best predictor of progression in PPMS

RESEARCH PLAN:

The investigators will enrol 30 primary-progressive MS subjects and 30 age- and sex-matched healthy controls to participate in two days of MRI experiments.

Whole-brain imaging will be performed on both days at Hvidovre Hospital on a research-only 7 Tesla Philips Achieva (Best, The Netherland) with a dual transmit, 32-channel receive head coil (Nova Medical).

Day 1: Submillimeter resolution anatomical images are collected for tissue segmentation, lesion identification, the assessment of central veins and paramagnetic rims.

In addition, a battery of physical and cognitive testing with a focus in sensorimotor hand function and cognitive processing speed will be performed, assessing two prominent symptoms of PPMS.

Day 2: Quantitative, spectroscopic (MRS) and functional MRI (fMRI) for the assessment of myelin.

ANALYSIS:

The main analysis will consist of cortical lesion identification, segmentation of both lesions and cortex and the assessment of the MRI myelin measures in both the lesions and NAGM. Control data will be used to establish a baseline measure of myelination. Myelin content in the different types of lesions and NAGM will be compared.

All statistical analysis will be performed in R. Linear and mixed effects modelling will determine how clinical, structural and MRI measures contribute to physical and cognitive performance, and will allow to extract the most relevant MR predictors of the clinical scores.

In part, the analysis will merge the acquired data with data from an ongoing study on structural and functional assessments for sensorimotor function in relapsing-remitting (RRMS) and secondary progressive MS (SPMS) (NCT03653585). This will allow to place the PPMS cohort directly in the context of other subtypes of MS.

The present study will significantly enhance the understanding of cortical damage in PPMS, the main contributor to chronic impairment. The non-invasive characterization of cortical lesions, structurally and in terms of myelin, will answer relevant questions about the brain's capacity for repair, the extent of demyelination and the occurrence of inherent cortical remyelination.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Diagnosed with primary progressive multiple sclerosis
* Expanded Disability Status Scale of ≤ 6.5
* No clinical relapse within last three months
* Have the ability to comply with all requirements of the study protocol, as determined by the investigator

Exclusion Criteria:

* Pregnancy
* Pacemaker or other implanted electronic devices
* Claustrophobia
* Psychiatric disorder
* Administration of acute cortisol
* Changes in pharmacological treatment within the last 3 months
* Any contraindication to MRI
* Persons who do not wish to be informed about abnormal findings as part of the investigations

HEALTHY CONTROLS

Inclusion Criteria:

* Able bodied
* Have the ability to comply with all requirements of the study protocol, as determined by the investigator

Exclusion Criteria:

* Pregnancy
* Under medication at the time of the experiment (with the exception of contraceptive drugs)
* History of neurologic disease
* Pacemaker or other implanted electronic devices
* History of cerebral hemorrhage or brain damage
* Claustrophobia
* Psychiatric disorder
* Any contraindication to MRI
* Persons who do not wish to be informed about abnormal findings as part of the investigations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy control volunteers will be recruited from the general population via the departments webpage (www.drcmr.dk), publicly available advertising media 'http://www.forsoegsperson.dk/', links on social media portal: 'facebook' and advertisements in newsstands and communication-boards in public facilities like canteens, educational institutions, sports facilities and hospitals in the Copenhagen area.
  Recruitment of 30 patients will be done through the ambulatory care at the Danish Multiple Sclerosis Center (DMSC) at Rigshospitalet in Copenhagen, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Distribution of cortical lesions in PPMS | Baseline
  Three different types of cortical lesions will be quantified across all cortical areas (Leuko- and Intracortical, Subpial). Their number in each area will be compared to existing data of RRMS and SPMS patients. Most patients are expected to show cortical lesions. It will be assessed which areas of the cortex are affected earliest in PPMS.
Volume of cortical lesions in PPMS | Baseline
  The volume of the different cortical lesion subtypes [in cubic mm] will be quantified and compared to lesion volumes in RRMS and SPMS patients. It will be assessed which type of damage, i.e. which of the three lesion types, drives motor and cognitive impairment using linear regression models. The investigators hypothesize that more extensive cortical demyelination will relate to lower/worse test scores.
Identify central veins and the presence of paramagnetic rims for cortical lesions | Baseline
  Susceptibility-sensitive imaging data will be pre-processed as described in literature and co-registered with other anatomical MRI data. It will be assessed whether the location of veins or paramagnetic rims matches areas of already identified lesions. Although central veins have gained large attention in white matter lesions as an additional diagnostic criterium, their presence and role in cortical lesions is less well understood. Paramagnetic rims of MS lesions have been identified as highly relevant predictors of active disease progression. Their prevalence in PPMS [in %] will be assessed and relationships to clinical, behavioural and MRI metrics will be explored in mixed effects models that account for other patients specific (age, gender, disease duration, EDSS) or lesion-specific variables (volume, lesion subtype).
Quantitative assessment of myelin density in cortical lesions, perilesional gray and white matter, and normal appearing cortex using myelin water imaging | Baseline
  On a group level, the myelin water fraction [in %] will be compared between cortical lesion subtypes and the normal appearing cortex. Lesions and normal appearing cortex are expected to have lower myelin density than cortical gray matter in non-neurological individuals. The variance in myelin density among lesions is expected to be high as various degrees of demyelination and remyelination may be present. Remyelination capacity of cortical lesions may be higher than in white matter lesions and thus myelin differences between cortical lesions and normal appearing cortex may be small. Myelin water fraction values will be assessed relative to clinical and behavioural metrics in mixed effects models. The investigators hypothesize that lower myelin densities, in addition to the volume of cortical demyelination, will relate to lower/worse test scores.
Quantitative assessment of magnetization transfer in cortical lesions, perilesional gray and white matter, and normal appearing cortex | Baseline
  Similarly, magnetization transfer indices will be assessed between lesion subtypes, normal appearing cortex and compared to cortical gray matter in non-neurological individuals. Instead of assessing directly the relaxation times of different water environments, MT provides an indirect assessment of the interaction of mobile and bound protons. Here, the macromolecular bound pool signal fraction [in %] will be assessed relative to clinical and behavioural metrics in mixed effects models. The investigators hypothesize that smaller pool fractions, in addition to the volume of cortical demyelination, will relate to lower/worse test scores.
Quantitative assessment of fractional anisotropy in cortical lesions, perilesional gray and white matter, and normal appearing cortex using diffusion tensor imaging data | Baseline
  Fractional anisotropy (FA) is a commonly used diffusion metric for the assessment of tightly packed, myelinated axons in white matter. FA and other diffusion metrics will be compared between the cortical lesion subtypes and the normal appearing cortex. On average, lower microstructural anisotropy is expected in lesions as a reflection of demyelination and partial axonal loss. FA values will be assessed relative to clinical and behavioural metrics in mixed effects models. The investigators hypothesize that lower FA, in addition to the volume of cortical demyelination, will relate to lower/worse test scores.

SECONDARY OUTCOMES:
Number of cortical lesions in the primary sensorimotor cortex (SM1) | Baseline
  Quantified as cortical lesion number on a unihemispheric level. The extent of damage to the SM1 is unknown, but based on clinical symptoms of motor function up to 40% of patients are expected to show focal cortical lesions in this area. The relationship between SM1 cortical lesion numbers and other MRI metrics (e.g. white matter lesion load of the corticospinal tract, cortical myelination, cortical thickness, metabolite levels of SM1-HAND and diffusion metrics of the corticospinal tract) will be assessed.
Cortical lesion volume in the primary sensorimotor cortex (SM1) | Baseline
  Cortical lesion volume is assessed on a unihemispheric level. Due to variable lesion size, the extent of damage to the SM1 may be better captured in terms of volume [cubic mm] than lesion number. The relationship between SM1 cortical lesion volume and other MRI metrics (e.g. white matter lesion load of the corticospinal tract, cortical myelination, cortical thickness, metabolite levels of SM1-HAND and diffusion metrics of the corticospinal tract) will be assessed.
Motor function | Baseline
  Upper and lower limb motor performance are assessed by 9-hole peg test and timed 25-foot walk. The investigators anticipate relationships of these scores with white matter integrity of motor tracts in the brain (corticospinal tract) and spinal cord cross sectional area (assessed on 3D MPRAGE data).
Sensory acuity | Baseline
  Sensory acuity is assessed as part of the EDSS on a scale between 1 and 5. The investigators anticipate relationships of these scores with white matter integrity of sensory tracts in the brain (corticospinal tract) and spinal cord cross sectional area (assessed on 3D MPRAGE data).
Regional metabolite concentration of the SM1 | Baseline
  Measured as N-acetylaspartate (NAA) concentration derived from MRS of a 2x2x2 voxel of the primary sensorimotor hand area. The NAA concentration within a lesioned hemisphere is expected to be decreased and to correlate with motor function, sensory acuity and regional myelin density. In addition, glutamate will be assessed, which is expected to be lower in PPMS than in HCs, and myo-inositol, which has been reported to be increased in RRMS compared to HCs. All metabolite concentrations are measured in [mM].
Functional MRI data for the assessment of temporal synchronization | Baseline
  A paradigm of finger movement paced by a visual cue will be used in a fMRI experiment to measure temporal synchronization as a proxy of sensorimotor organization and cortical myelination. The investigators anticipate reduced synchronization with higher EDSS and lower myelin density.
Cognitive performance and relationship to MRI measures (Exploratory) | Baseline
  Cognitive performance related to information processing speed and encoding, recall and recognition is assessed using the symbol digit modalities test (SDMT) and the California Verbal Learning Test (CVLT II). In an exploratory analysis, it will be assessed if cognitive performance scores relate to myelin changes in specific areas of the brain, both in gray and white matter, and whether there is a relationship with cortical lesion load.

OTHER OUTCOMES:
Depression | Baseline
  Depression score from the Beck depression inventory II (BDI-II) questionnaire (range 0-63, lower being less depressed).
Fatigue | Baseline
  Fatigue will be assessed using the Fatigue Scale for Motor and Cognitive Functions (FSMC), 20 item questionnaire (10 motor, 10 cognitive items) with each item's response rated on a 5-point Likert scale. Lower scores indicate less fatigue.
Morphometric measures: Whole brain cortical volume and white matter lesion volume (covariate) | Baseline
  Volume of cortical gray matter and white matter lesion volume [cubic mm] derived from segmented MR images.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Wiggermann, PhD, Principal Investigator — Danish Research Centre for Magnetic Resonance; Hartwig R Siebner, Prof, Study Director — Danish Research Centre for Magnetic Resonance
Locations (1):
- Danish Research Centre for Magnetic Resonance, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
In accordance with Danish data protection legislation, it is currently not allowed to publish individual participant data.
  Data that underlie published results related to the primary and secondary outcome measures will, following anonymization, be made publicly available. However, data will be grouped in appropriate age categories with minimum 5 participants in each group.

REFERENCES:
- [Background] Miller DH, Leary SM. Primary-progressive multiple sclerosis. Lancet Neurol. 2007 Oct;6(10):903-12. doi: 10.1016/S1474-4422(07)70243-0. PMID 17884680
- [Background] Nielsen AS, Kinkel RP, Madigan N, Tinelli E, Benner T, Mainero C. Contribution of cortical lesion subtypes at 7T MRI to physical and cognitive performance in MS. Neurology. 2013 Aug 13;81(7):641-9. doi: 10.1212/WNL.0b013e3182a08ce8. Epub 2013 Jul 17. PMID 23864311
- [Background] Cocozza S, Cosottini M, Signori A, Fleysher L, El Mendili MM, Lublin F, Inglese M, Roccatagliata L. A clinically feasible 7-Tesla protocol for the identification of cortical lesions in Multiple Sclerosis. Eur Radiol. 2020 Aug;30(8):4586-4594. doi: 10.1007/s00330-020-06803-y. Epub 2020 Mar 24. PMID 32211962
- [Background] Louapre C, Govindarajan ST, Gianni C, Langkammer C, Sloane JA, Kinkel RP, Mainero C. Beyond focal cortical lesions in MS: An in vivo quantitative and spatial imaging study at 7T. Neurology. 2015 Nov 10;85(19):1702-9. doi: 10.1212/WNL.0000000000002106. Epub 2015 Oct 14. PMID 26468411
- [Background] Kutzelnigg A, Lucchinetti CF, Stadelmann C, Bruck W, Rauschka H, Bergmann M, Schmidbauer M, Parisi JE, Lassmann H. Cortical demyelination and diffuse white matter injury in multiple sclerosis. Brain. 2005 Nov;128(Pt 11):2705-12. doi: 10.1093/brain/awh641. Epub 2005 Oct 17. PMID 16230320
- [Background] Chang A, Staugaitis SM, Dutta R, Batt CE, Easley KE, Chomyk AM, Yong VW, Fox RJ, Kidd GJ, Trapp BD. Cortical remyelination: a new target for repair therapies in multiple sclerosis. Ann Neurol. 2012 Dec;72(6):918-26. doi: 10.1002/ana.23693. Epub 2012 Oct 17. PMID 23076662
- [Background] Absinta M, Sati P, Schindler M, Leibovitch EC, Ohayon J, Wu T, Meani A, Filippi M, Jacobson S, Cortese IC, Reich DS. Persistent 7-tesla phase rim predicts poor outcome in new multiple sclerosis patient lesions. J Clin Invest. 2016 Jul 1;126(7):2597-609. doi: 10.1172/JCI86198. Epub 2016 Jun 6. PMID 27270171
- [Background] MacKay A, Whittall K, Adler J, Li D, Paty D, Graeb D. In vivo visualization of myelin water in brain by magnetic resonance. Magn Reson Med. 1994 Jun;31(6):673-7. doi: 10.1002/mrm.1910310614. PMID 8057820
- [Background] Ingle GT, Thompson AJ, Miller DH. Magnetic resonance imaging in primary progressive multiple sclerosis. J Rehabil Res Dev. 2002 Mar-Apr;39(2):261-71. PMID 12051469
- [Background] Dal-Bianco A, Grabner G, Kronnerwetter C, Weber M, Hoftberger R, Berger T, Auff E, Leutmezer F, Trattnig S, Lassmann H, Bagnato F, Hametner S. Slow expansion of multiple sclerosis iron rim lesions: pathology and 7 T magnetic resonance imaging. Acta Neuropathol. 2017 Jan;133(1):25-42. doi: 10.1007/s00401-016-1636-z. Epub 2016 Oct 27. PMID 27796537
- [Background] Wiggermann V, MacKay AL, Rauscher A, Helms G. In vivo investigation of the multi-exponential T2 decay in human white matter at 7 T: Implications for myelin water imaging at UHF. NMR Biomed. 2021 Feb;34(2):e4429. doi: 10.1002/nbm.4429. Epub 2020 Oct 28. PMID 33118238